CLINICAL TRIAL: NCT00480987
Title: A Phase I-II Study of Oxaliplatin, Fludarabine, and Cytarabine in Patients With Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndromes at First Relapse With Complete Remission Duration < 1 Year
Brief Title: Oxaliplatin, Fludarabine, and Cytarabine in Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of support.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-1089
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Leukemia
Keywords: High-Risk Myelodysplastic Syndromes; Acute Myeloid Leukemia; Leukemia; Oxaliplatin; Fludarabine; Cytarabine; AML; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia | interventions — Oxaliplatin; fludarabine; fludarabine phosphate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin + Cytarabine + Fludarabine (Experimental): Oxaliplatin 30 mg/m^2 intravenous (IV) days 1-4, Cytarabine 500 mg/m^2 by IV continuous infusion days 2-6, Fludarabine 30 mg/m^2 IV days 2-6
  Interventions: Drug: Oxaliplatin; Drug: Fludarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Oxaliplatin — 30 mg/m^2 IV days 1-4
  Other Names: Eloxatin®
Drug: Fludarabine — 30 mg/m^2 IV days 2-6
  Other Names: Fludara®; Fludarabine Phosphate
Drug: Cytarabine — 500 mg/m^2 by IV continuous infusion days 2-6
  Other Names: Ara-C

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of oxaliplatin combined with fludarabine plus cytarabine that can be given to patients with Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndromes (MDS). Once the highest tolerable dose of oxaliplatin in this drug combination is found, the next goal of the study will be to learn the safety and the ability of the drug combination to control the disease.

DETAILED DESCRIPTION:
The Study Drugs:

Cytarabine is designed to insert itself into Deoxyribonucleic acid (DNA) (the genetic material of cells) and stop the DNA from repairing itself.

Fludarabine is designed to make cancer cells less able to repair damaged DNA. This may increase the likelihood of the cells dying.

Oxaliplatin is designed to "program" cells to cause death in leukemic cells.

The Phases of The Study:

This research study has 2 parts, Phase I and Phase II.

The Phase I part of the study will be used to test different dose levels in order to determine the highest tolerable dose of the study drug oxaliplatin that can be given in combination with cytarabine and fludarabine to patients with AML or high-risk MDS. Three (3) participants will be enrolled at each dose level until the highest tolerable dose is found.

The Phase II part of the study will evaluate the safety and disease-control ability of the study drug combination (the highest tolerable dose that was found) in order to treat these patients.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will be given oxaliplatin through a needle (intravenously -- through an IV) in your vein over 2 hours for 4 days (Days 1-4) in a row.

On Day 2, you will be given cytarabine through an IV in your vein by continuous infusion over 24 hours for 5 days (Days 2-6) in a row. Starting on Day 2, you will be given fludarabine through an IV in your vein over 30 minutes for 5 days (Days 2-6) in a row. In order to keep you from being dehydrated, you will also be given other IV fluids, such as saline (a salt solution), each day you receive the study drugs. If the drugs are given on an outpatient basis, a daily visit may take about 8 hours.

One (1) cycle is 6 days long. The first cycle will be given at M. D. Anderson. Each cycle will be repeated every 4-6 weeks. Depending on your response to the study drug combination, you will have up to 5 more cycles either at M. D. Anderson or on an outpatient basis with your regular physician.

Your study drug dose may be lowered if you experience severe side effects.

Study Visits:

During each treatment cycle, you will have blood drawn (about 1 teaspoon each time) at least 2-3 times a week for routine tests. You will have a bone marrow aspiration done on Day 21 of Cycle 1 and once a week thereafter, unless there is clear evidence of active disease. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

Length of Study:

You will remain on this study for up to 6 cycles for a total of about 6 months, unless the disease is not responding, the disease gets worse, or you experience intolerable side effects. If you are taken off this study early, your study doctor will discuss other treatment options with you.

End-of-Treatment Visit:

Once you have completed treatment on this study, you will have an end-of-treatment visit. This visit will include routine blood tests (about 1 teaspoon will be drawn each time) and a bone marrow aspirate to check the status of the disease. If your blood tests show the disease has gotten worse, no bone marrow aspirate will be needed.

Long-Term Follow-up:

After your last cycle of treatment is completed and every 3 months for as long as you are in remission, you will have blood drawn (about 2 teaspoons each) for routine testing.

This is an investigational study. Cytarabine is Food and Drug Administration (FDA) approved and commercially available for the treatment of AML and other blood cancers. Fludarabine is FDA approved and commercially available for the treatment of chronic lymphocytic leukemia (CLL). Oxaliplatin is FDA approved and commercially available for the treatment of advanced colorectal cancer and colon cancer. Their use in combination is investigational in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed relapsed or refractory acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome.
* Performance status 0-2 (Zubrod scale).
* Serum creatinine equal or less than 1.3 mg/dL or creatinine clearance > 40 mL/min.
* Bilirubin </= 2 mg/dL; serum glutamic oxaloacetic transaminase (SGOT) or Serum glutamic pyruvic transaminase (SGPT) </= 3 times the Upper Limit of Normal (ULN) for the reference lab unless due to leukemia or congenital hemolytic disorder (for bilirubin).
* Written informed consent.

Exclusion Criteria:

* No untreated or uncontrolled life-threatening infection.
* No oxaliplatin, fludarabine, or cytarabine intolerance.
* No pregnancy or lactation. Female patients of childbearing potential (including those < 1 year post-menopausal) and male patients must agree to use contraception.
* No chemotherapy or radiation therapy within 4 weeks of study entry. Hydroxyurea is allowed prior to starting therapy in the setting of rapidly proliferating disease.
* No other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent or cooperate and participate in the study or to interfere with the interpretation of the results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 1/15/08 - 11/3/09; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: There were 27 participants registered and all were included in the analysis. The trial terminated early.
Period: Overall Study
Arm/Group | Oxaliplatin + Cytarabine + Fludarabine
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin + Cytarabine + Fludarabine
Number analyzed (Participants) | 27
Age Continuous [Median (Full Range); unit: years] | 58 [6 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response: Complete Response/Remission (CR) defined as a bone marrow with 5% or fewer blasts and peripheral blood count with an absolute neutrophil count of 10^9/Liters or more and platelet count of 100*10^9/Liters or more; Complete Response with Platelets/remission without platelet recovery (CRp) defined as a complete response except for a platelet less than 100*10^9/Liters and transfusion independent; and Partial Response/Remission defined as peripheral blood count recovery as for CR with decrease in marrow blasts >/= 50% and not more than 6-25% abnormal cells in the marrow.
Time Frame: After 2 months
Population: Analysis was per protocol. All participants treated were analyzed.
Measure: Number; unit: Participants
Arm/Group | Oxaliplatin + Cytarabine + Fludarabine
Number analyzed (Participants) | 27
Participants
  Complete response | 3
  Complete response with platelets | 2
  Partial response | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Oxaliplatin + Cytarabine + Fludarabine
Serious Adverse Events (participants affected / at risk) | 5/27
Other Adverse Events (participants affected / at risk) | 10/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin + Cytarabine + Fludarabine (N=27)
Pneumonia (Infections and infestations) | 2 (2)
Death (General disorders) | 5 (5) — Disease Progression
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin + Cytarabine + Fludarabine (N=27)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Hyperbilirubinemia (Hepatobiliary disorders) | 3 (3)
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes